CLINICAL TRIAL: NCT06199960
Title: Comparison of Two Types of Dual Ovarian Stimulation: Duostim Versus Shanghai Protocols in Patients With Poor Ovarian Reserve: A Randomized Controlled Trial
Brief Title: Dual Ovarian Stimulation (Duostim) and Shanghai Protocols in Poor Ovarian Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97000185
Record Dates: First submitted 2021-02-09; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Assisted Reproductive Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double GnRH-antagonist protocol (Duostim protocol) (Experimental): In Duostim group, both follicular and luteal phases stimulation will perform with 150-225 IU of recombinant FSH (Gonal-F®, Merck-sereno, Germany) and HMG (Humegnan, Darou Pakhsh Co., Iran) in GnRH antagonist treatment. The follicular stimulation will be started on day 2-3 of the menstrual. Daily administration of 0.25 mg of GnRH antagonist (Cetrotide®, Merck-Serono; Germany) will be started when the leading follicle are 13-14mm and continue until the day of the oocyte trigger. When one follicle reached 17-18 mm ovulation will be triggered with 0.5 cc of Buserelin acetate (CinnaFact®; CinnaGen pharmaceutical Co., Iran) and oocyte retrieval will be performed after 34-36 hours. Five days after the ﬁrst oocyte retrieval, a GnRH antagonist protocol identical to the ﬁrst one will start. When at least two follicles reached 17-18 mm, the ovulation will be triggered with a subcutaneous bolus GnRH-agonist and the second oocyte retrieval will be performed.
  Interventions: Other: Doustim protocol
- Double mild stimulation protocol (No Intervention): In double mild stimulation protocol, Clomiphene citrate 25 mg/day (Ovumid®; Iran Hormone pharmaceutical Co., Iran) and co-treatment with letrozole 2.5 mg/day (Femati®, Atipharmed Co., Iran) will be given from cycle day 3. Letrozole is given for 4 days and clomiphene citrate is used daily before the trigger day. Patients take 150 IU of Human menopausal gonadotropin (HMG) (Humegnan®, Darou Pakhsh Co., Iran) every other day beginning on cycle day 6. When one dominant follicle will reach 18 mm, the ﬁnal triggering will induce 34-36 h after 0.5 cc of Buserelin acetate (CinnaFact®; CinnaGen pharmaceutical Co., Iran) administration. In luteal phase stimulation a total of 225 IU HMG and letrozole 2.5 mg will administered daily from3 to 5 days after oocyte retrieval. Letrozole administration will be stopped when the dominant follicles reached 12 mm. When one dominant follicle will reach 18 mm, the ﬁnal triggering will be induced with 0.5 cc of Buserelin acetate.

INTERVENTIONS:
Other: Doustim protocol — In Duostim group, the follicular stimulation will be started with a ﬁxed dose of 150 IU of rFSH and HMG 75 IU for 4 days. Daily administration of a GnRH antagonist will be started when the leading follicle are 13-14mm in diameter and continue until the day of the trigger of the ovulation. Five days after the ﬁrst oocyte retrieval second gonadotropin stimulation will be started identical to the ﬁrst one..
  Other Names: Double GnRH-antagonist stimulation
  Arms: Double GnRH-antagonist protocol (Duostim protocol)

SUMMARY:
A combination of follicular phase stimulation and luteal phase stimulation in the same cycle, can be a valuable choice in poor responder patients with reduced ovarian reserve, in order to achieve extreme the number of oocytes in a single menstrual cycle. In the present study, the results of two different Double stimulation cycles including shanghai protocol and Duostim protocol in patients with reduced ovarian reserve, compared with each other to help select a more appropriate treatment for this group of patients. The number of retrieved oocytes and the number of obtained embryos and clinical pregnancy from each protocol will be compared as the primary and secondary outcome.

DETAILED DESCRIPTION:
The proposal of this randomized clinical trial study is a comparison of two different type of double stimulation protocols in patients who meet the POSEIDON (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number) stratification (group 4) criteria.

In mild double stimualtion (Shanghai protocol), patients will be received Clomiphene citrate 25 mg/day (Ovumid®; Iran Hormone pharmaceutical Co., Iran) co-treatment and letrozole 2.5 mg/day (Femati®, Atipharmed Co., Iran) will be given from cycle day 3. Letrozole is given for 4 days and clomiphene citrate is used daily before the trigger day. Patients take 150 IU of Human menopausal gonadotropin (HMG) (Humegnan®, Darou Pakhsh Co., Iran) every other day beginning on cycle day 6. When one dominant follicle will reach 18 mm, the ﬁnal triggering will induce 34-36 h after 0.5 cc of Buserelin acetate (CinnaFact®; CinnaGen pharmaceutical Co., Iran) administration. In luteal phase stimulation a total of 225 IU HMG and letrozole 2.5 mg will administered daily from3 to 5 days after oocyte retrieval. Letrozole administration will be stopped when the dominant follicles reached 12 mm. When one dominant follicle will reach 18 mm, the ﬁnal triggering will be induced with 0.5 cc of Buserelin acetate (CinnaFact®; CinnaGen pharmaceutical Co., Iran).

In the double GnRH- antagonist (Duostim protocol), both follicular and luteal phases stimulation will perform with 150-225 IU of recombinant FSH (Gonal-F®, Merck-sereno, Germany) and HMG (Humegnan, Darou Pakhsh Co., Iran) in GnRH antagonist treatment. The follicular stimulation will be started on day 2-3 of the menstrual. Daily administration of 0.25 mg of GnRH antagonist (Cetrotide®, Merck-Serono; Germany) will be started when the leading follicle are 13-14mm and continue until the day of the oocyte trigger. When one follicle reached 17-18 mm ovulation will be triggered with 0.5 cc of Buserelin acetate (CinnaFact®; CinnaGen pharmaceutical Co., Iran) and oocyte retrieval will be performed after 34-36 hours. Five days after the ﬁrst oocyte retrieval, a GnRH antagonist protocol identical to the ﬁrst one will start. When at least two follicles reached 17-18 mm, the ovulation will be triggered with a subcutaneous bolus GnRH-agonist and the second oocyte retrieval will be performed.

In all of groups all of embryos will be freeze and will be used in subsequent frozen embryo transfer (FET) cycles. Endometrial preparation for FET cycle will perform with hormonal replacement therapy (HRT) cycle protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥35 years
2. Antimullerian hormone (AMH) <1.2 ng/ml and/or Antral follicular count≤5 follicles
3. ≤4 oocyte retrieved from previous ART cycle 4-18.5<BMI<30

Exclusion Criteria:

1. Endometriosis (stage III and IV)
2. Myoma with a compression effect
3. Uterine anomalies (Unicorn, Didelphis,etc,….)
4. Male factor infertility with azoospermia, severe oligospermia and oligoasthenospermia, TESE/PESA

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Number of MII oocytes | Immediately after oocyte puncture
  Oocytes that were mature at the time of oocyte collection (Metaphase II)

SECONDARY OUTCOMES:
Number of cleaved embryos | 2-3 days after oocyte puncture
  2-3 days embryo from fertilization
Number of blastocyst embryos | 5 days after oocyte puncture and sperm insemination
  The stage the embryo reaches after 5 days in culture from the oocyte retrieval
Clinical pregnancy rate | 4-6 weeks after embryo transfer
  The observation of gestational sac on ultrasound examination two-three weeks after positive serum βhCG
Fertilization rate | 2-5 days after sperm insemination
  Percentage of transformation of micro injected oocytes into two pronuclei
Quality of oocytes | Immediately after oocyte puncture
  Oocyte quality were assessed by embryologist based on The Istanbul consensus workshop (Hum Reprod.2011). Quality of MII oocytes (based on intracytoplasmic and extracytoplasmic abnormalities) was divided into 3 groups; morph, slightly dysmorph, and dysmorph.

CONTACTS AND LOCATIONS:
Overall Officials: Mehri Mashayekhi, M.D, Principal Investigator — Department of Endocrinology and Female Infertility
Locations (1):
- Royan Institute, Tehran, Iran